CLINICAL TRIAL: NCT02900456
Title: The Intra-Aortic Balloon Pumps Insertion Registry on Behalf of the Groupe Des Angioplasticiens de la Région Ouest
Acronym: CP-GARO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_8942
Record Dates: First submitted 2016-08-26; First posted 2016-09-14 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Interventional Cardiology
Keywords: Intra-aortic Balloon Pumps; Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Intra-aortic Balloon Pumps (IABP) have been used for roughly 50 years in Critical Care Units, Intensive Care Units, Cath labs as a way to improve systemic and coronary circulation in patients in cardiogenic shock (CS) or at high risk situation as mechanical complications stemming from myocardial infarction (MI), critical coronary stenosis, high-risk PCI, etc. Several papers recently questioned the relevance of this assistance device - namely the IABP-SHOCK II trial in CS and the CRISP-AMI trial in anterior MI without CS - resulting in the downgrading of the recommendation standards of the IABP by medical societies.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least of 18 of age;
* Undergoing IABP treatment ;
* Subject, relatives or legal guardian signified their non-opposition to participate in the study

Exclusion Criteria:

- IABP insertion in immediate post-intervention period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intra-aortic Balloon Pumps in patients in cardiogenic shock (CS) or at high risk situation as mechanical complications stemming from myocardial infarction (MI), critical coronary stenosis, high-risk PCI, etc
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
IABP insertion rate | 1 year

SECONDARY OUTCOMES:
Number of cardiogenic shock | 1 year
  IABP indications
Number of mechanical complication of acute coronary syndrome | 1 year
  IABP indications
Number of myocardial infarction not shocked | 1 year
  IABP indications
Number of other indications | 1 year
  IABP indications
Survival rate following IABP insertion | 1 year
IABP-related complications rate and type | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEURENT, Principal Investigator — CHU Rennes
Locations (25):
- France (25):
  - CHU Angers, Angers
  - Clinique Saint Joseph, Angers
  - CHU Brest, Brest
  - CHU Caen, Caen
  - Hôpital Prive Saint Martin, Caen
  - CH Chartres, Chartres
  - CH Laval, Laval
  - CH Le Mans, Le Mans
  - CH Bretagne Sud, Lorient
  - CHU Nantes, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CH Intercommunal de Cornouaille, Quimper
  - CHU Rennes, Rennes
  - Hôpital privé Beauregard, Rennes
  - Polyclinique Saint-Laurent, Rennes
  - CHU Rouen, Rouen
  - Clinique Saint-Hilaire, Rouen
  - CH Saint-Brieuc, Saint-Brieuc
  - CH Saint-Nazaire, Saint-Nazaire
  - Groupement Coopération Sanitaire Pui Cite Sanitaire, Saint-Nazaire
  - Communauté Hospitalière de Territoire Rance Emeraude, St-Malo
  - Polyclinique Les Fleurs, Toulon
  - CHU Tours, Tours
  - Clinique Saint Gatien, Tours
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No